CLINICAL TRIAL: NCT01697280
Title: Improving Routine Immunization Coverage Through Educational Messages Delivered During Polio NIDs in Pakistan: A Cluster Randomized Trial
Brief Title: Polio NID and Routine EPI Integration Trial Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Principal Investigator, Anita Kaniz Mehdi Zaidi, Professor and Chair, Department of Paediatrics and Child Health, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1952-Ped-ERC-11
Record Dates: First submitted 2012-04-02; First posted 2012-10-02 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Polio
Keywords: Polio supplementary immunization activities; Routine EPI vaccine; Integration of polio NID and routine EPI
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Educational messages only (Experimental): EPI vaccinators/volunteers will educate mothers/care-providers of infants less than 12 months old months about the benefits of routine immunization
  Interventions: Behavioral: Vaccine promotion messages; Other: Distribution of Plastic Pouches to retain vaccination card
- Immunization status verification only (Experimental): EPI vaccinators/volunteers will identify and record details of un/under-vaccinated children less than 12 months old in households they visit during an NID, and update immunization registries maintained at the local EPI centers so these children can be reached in subsequent outreach activity.
  Interventions: Other: Vaccination Verification.; Other: Distribution of Plastic Pouches to retain vaccination card
- Education and vaccine verification (Experimental): EPI vaccinators/volunteers will educate mothers/care-providers of infants less than 12 months old months about the benefits of routine immunization, identify and record details of un/under-vaccinated children in households they visit during an NID, and update immunization registries maintained at the local EPI centers so these children can be reached in subsequent outreach activity.
  Interventions: Behavioral: Vaccine promotion messages; Other: Vaccination Verification.; Other: Distribution of Plastic Pouches to retain vaccination card
- Status quo (No Intervention): No interventional activity will take place in this group. Therefore, the status quo (routine services) will be maintained during Polio NID

INTERVENTIONS:
Behavioral: Vaccine promotion messages — The messages will be low-literacy, of very short duration, and will be delivered with the help of pictorial cards. These educational messages will include the following messages:
  1. Vaccines can save a child's life
  2. Children who are immunized on time are less likely to become ill
  3. Unimmunized children can become disabled for life
  4. Photograph of the nearest EPI center where vaccines are offered free of charge, as well as its address and timings.
  Arms: Education and vaccine verification; Educational messages only
Other: Vaccination Verification. — EPI vaccinators/volunteers will identify and record details of un/under-vaccinated children less than 12 months old in households they visit during an NID, and update immunization registries maintained at the local EPI centers so these children can be reached in subsequent outreach activity.
  Arms: Education and vaccine verification; Immunization status verification only
Other: Distribution of Plastic Pouches to retain vaccination card — At the start of this project, all EPI centers in the study areas will be provided with plastic pouches to be given to parents of all children coming to EPI centers for vaccinations. These pouches will be used to store a child's immunization card.
  Arms: Education and vaccine verification; Educational messages only; Immunization status verification only

SUMMARY:
This study aims to assess if pictorial messages promoting routine immunization during supplementary campaigns for oral polio vaccine in areas with poor DTP3 vaccine coverage can improve immunization rates. A cluster randomized trial design in low literature populations will be used.

DETAILED DESCRIPTION:
The overall objective of this study is to assess whether supplementary immunization activities (SIAs) held for polio eradication can be used to improve routine immunization coverage in Pakistan.

Primary research objectives:

(i) To assess effectiveness of educational messages regarding routine immunization during SIAs held for polio on improving routine immunization coverage in Pakistan.

Secondary research objectives:

(i) To assess maternal knowledge about routine immunization in the intervention and control arms.

(ii) To estimate vaccination card retention in the intervention and control arms.

This study will be completed in 12 months, between March 2012 to February 2013. Overall, three major operational steps have been defined for the study as follow:

Baseline vaccine coverage survey: This is a 02-months activity in which a baseline household vaccine coverage survey will be carried out to independently assess the immunization coverage and socio-demographic indicators in the study areas. Participation in this survey will be voluntary and written consent from participants will be obtained prior to administering the study questionnaire.

Training of vaccinators/volunteers and distribution of plastic pouches: The project research staff (Research Associate/Senior Research Assistants) will be exclusively trained by Principal Investigator/Research Supervisor on educational material. Having completed the baseline coverage survey, a one-day training session will be organized by trained project staff to provide trainings to participating EPI vaccinators/volunteers on the vaccine promotion educational messages to be delivered during intervention. These trainings will be held at a common venue (EPI center/public hospital) in the selected towns for this study. The messages will be low-literacy, of very short duration, and will be delivered with the help of pictorial cards which were previously developed for and used in a similar department-run study in Karachi. These educational messages will include the following messages:

1. Vaccines can save a child's life
2. Children who are immunized on time are less likely to become ill
3. Unimmunized children can become disabled for life
4. Photograph of the nearest EPI center where vaccines are offered free of charge, as well as its address and timings

Additionally, at the start of this project, all EPI centers in the study areas will be provided with plastic pouches to be given to parents of all children coming to EPI centers for vaccinations. These pouches will be used to store a child's immunization card. In order to assess the likely change in vaccination card retention, we will compare the proportion of vaccination cards available on pre-and-post coverage assessment in both intervention and control groups.

Endline vaccine coverage survey/outcome assessment. Outcome assessment will be done through a representative endline survey assessing vaccine coverage for Penta-3 and Measles-1 in the study areas, 3 months after the NID was held. Participation in this survey will be voluntary and written consent from study participants will be obtained prior too administering the study questionnaire.

NID = National Immunization Days SNID = Sub-national Immunization Days EPI: Expanded Programme on Immunization SIA - Supplementary Immunization Activity CHW = Community Health Worker AKU = Aga Khan University, Karachi, Pakistan

ELIGIBILITY:
Inclusion Criteria:

1. Households with children aged 3-14 months
2. Resident of selected cluster
3. Willing to consent for participation in the study

Exclusion Criteria:

1. Households with children aged below 3 months or above 14 months
2. Non-resident of selected cluster
3. Refusing to consent

Ages: 3 Months to 14 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4560 (Actual)
Dates: Start 2012-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
age appropriate vaccination of children 3 - 14 months old at the time of the endline survey | 03 months after intervention (polio NID)
  Age appropriate vaccination for the purposes of this study is defined as the administration of:
  1. All scheduled doses of the DPT/Hepatitis-B/Hib (Penta) vaccine within 14 days of the recommended age for children 3 - 11 months of age, and
  2. First dose of the measles vaccine (Measles-1) for children 9 - 14 months of age.

SECONDARY OUTCOMES:
Maternal knowledge about routine immunization | 03 months after intervention
  Maternal knowledge about nearest EPI facility, names of EPI vaccines that child is age-eligible to receive, cost of vaccination and importance about vaccination will be assessed during end line vaccine coverage survey.
Retention of immunization cards | 03 months after intervention (polio NID)
  The number of children who received routine EPI vaccine had vaccination card available on the end-line survey. Immunization cards will help to verify dates and number of doses that child has received.

CONTACTS AND LOCATIONS:
Overall Officials: Anita KM Zaidi, MBBS, FAAP, Principal Investigator — Aga Khan University
Locations (1):
- Thatta, Hyderabad, Thatta, Hyderabad, Sindh, Pakistan